CLINICAL TRIAL: NCT00255866
Title: Improving Affect and Behavior in Assisted Living Residents
Brief Title: Improving Mood and Behavior in Assisted Living Residents Through Skills Training for Their Caregivers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linda Teri, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 26082-ED; R21MH069651 (NIH); DSIR 82-SEDR
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-12

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Assisted Living Facilities; Aged; Elderly; Caregivers
MeSH Terms: conditions — Dementia; Alzheimer Disease

INTERVENTIONS:
Behavioral: Skills training for the care of dementia patients

SUMMARY:
This study will develop a treatment program to reduce mood and behavior problems in assisted living residents who have dementia.

DETAILED DESCRIPTION:
Assisted living is rapidly becoming one of the most common methods of caring for older adults with dementia in long-term care. Over half of assisted living residents have dementia and many exhibit affective and behavioral problems related to the condition; residents' care and quality of life may suffer as a result of these problems. Despite the seriousness of this condition, interventions to teach direct care staff how to care for these residents are limited. This study will develop a program for teaching assisted living staff how to deal with the issues of patients with dementia and reduce mood and behavioral problems among this population.

Caregivers will be randomly assigned to attend skills training sessions as two 4-hour workshops, four 30 minute individual training sessions, or two 30 minute in-services. Training will focus on dementia, depression and anxiety, the incidence of behavior problems, and skills and techniques for alleviating care challenges associated with behavior problems. Caregivers will complete self-report scales and questionnaires at the beginning and at the end of the study; these measures will assess job satisfaction, reactions to resident behavioral problems, and job skills. Residents will also be recruited for this study; they will complete questionnaires about their depressive episodes, anxiety, behavioral problems, and quality of life at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria for Assisted Living Staff

* Work in the assisted living residence for at least 6 months prior to study entry
* Work in the assisted living residence at least 5 days a week, for at least 4 hours a day on day or afternoon-evening shifts
* Provide direct care for at least 1 assisted living resident
* Agree to attend all training sessions and complete assessment forms
* Able to speak, read, and understand English at a 6th grade level

Inclusion Criteria for Assisted Living Residents:

* Diagnosis of dementia
* Identified by caregiving staff as having mood or behavioral problems
* Have lived at the assisted living residence for at least 3 months prior to study entry
* Have a family member with power of attorney

Exclusion Criteria for Assisted Living Residents:

* Plan to receive medication for affective or behavioral problems during the study
* History of alcohol or drug abuse
* Have attempted suicide within 1 year prior to study entry

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Skills to effectively deal with resident behavioral problems

SECONDARY OUTCOMES:
Resident depression, anxiety, behavioral problems, and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Linda Teri, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Rush University School of Nursing, Chicago, Illinois